CLINICAL TRIAL: NCT00299481
Title: Tissue and Data Acquisition Activity for the Study of Gynecological Disease
Brief Title: Tissue Bank of Biological Specimens From Patients With Gynecologic Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Collaborators: Walter Reed Army Medical Center (U.S. Federal Agency); Ohio State University (Other); University of Pittsburgh (Other); Duke University (Other); H. Lee Moffitt Cancer Center and Research Institute (Other); Windber Research Institute (Other); Medstar Health Research Institute (Other)
Organization: Walter Reed Army Medical Center (U.S. Federal Agency)
Other Study IDs: 04-44017; W81XWH-05-2-0005; A-12818.1a
Record Dates: First submitted 2006-03-02; First posted 2006-03-06 (Estimated); Last update posted 2008-06-30 (Estimated); Status verified 2008-06

CONDITIONS: Endometrial Neoplasms; Uterine Cervical Neoplasms; Ovarian Neoplasms; Leiomyoma
Keywords: Tissue Bank; Endometrial neoplasm; uterine cervical neoplasm; ovarian neoplasm; leiomyoma; DNA; RNA; Protein; Serum
MeSH Terms: conditions — Endometrial Neoplasms; Uterine Cervical Neoplasms; Ovarian Neoplasms; Leiomyoma

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
The purpose of this study is to create a tissue bank of gynecologic cancers and normal tissue for the study of cancer in order to better understand the changes occurring on a molecular level (DNA, RNA, protein) that lead to the development of cancer.

DETAILED DESCRIPTION:
Cancer arises due to genetic alterations that disrupt numerous cellular functions including proliferation, programmed cell death and senescence, that ultimately control the number of cells in a population. The genetic damage that underlies the development of cancers has a diverse etiology and loss of DNA repair mechanisms also may play a role in allowing mutations to accumulate. Cancers are also characterized by the ability to invade surrounding tissues and to metastasize. Many of the molecular alterations involved in this process have yet to be elucidated.

Gynecologic cancers afflict women of all ages. Cervical cancer is the most common gynecologic malignancy worldwide, accounting for over 400,000 cases annually. Endometrial cancer is the most common gynecologic malignancy with approximately 33,000 new cases being diagnosed annually in American women. Ovarian cancer is the fourth most common cause of cancer related mortality in American women, with approximately 14,000 deaths occurring from it in 2000.

The creation of a tissue repository containing tissue specimens, blood/serum, and molecular extracts (DNA, RNA, protein) will provide a rich source of tissue for future gynecological disease research studies.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled to undergo surgery for diagnosis and treatment of a gynecologic disease at one of the participating institutions
* > = 18 years old
* Ability to read English

Exclusion Criteria:

* < 18 years old

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7000 (Estimated)
Dates: Start 2006-03; Study Completion 2011-01

CONTACTS AND LOCATIONS:
Overall Officials: LTC G. Larry Maxwell, MD, Principal Investigator — Walter Reed Army Medical Center
Locations (7):
- United States (7):
  - Washington Hospital Center, Washington D.C., District of Columbia
  - Gynecologic Disease Center, Walter Reed Army Medical Center, Washington D.C., District of Columbia
  - Wayne State University Kamanos Cancer Institute, Detroit, Michigan
  - Duke University Medical Center, Durham, North Carolina
  - The Ohio State University, Columbus, Ohio
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Windber Research Institute, Windber, Pennsylvania